CLINICAL TRIAL: NCT01611831
Title: Efficacy of Acceptance and Commitment Therapy (ACT) in Group in Fibromyalgia: a Randomized, Controlled Study.
Brief Title: Efficacy of Acceptance and Commitment Therapy (ACT) in Group in Fibromyalgia
Acronym: ACTGROUP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dr. Marta Alda (Other)
Collaborators: Instituto Aragones de Ciencias de la Salud (Other Government); Carlos III Health Institute (Other Government)
Responsible Party: Sponsor-Investigator, Dr. Marta Alda, Principal Investigator, Hospital Miguel Servet
Organization: Hospital Miguel Servet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI11/024
Record Dates: First submitted 2012-05-11; First posted 2012-06-05 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-05

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; Acceptation & Commitment Therapy; randomized controlled trial
MeSH Terms: conditions — Fibromyalgia | interventions — Population Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ACT in group (Experimental): Patients assigned to this arm will receive Acceptation and Commitment Therapy (ACT) in groups of 8-12 patients. Intervention has been protocolized. Therapy will be administered by two experienced therapists (psychologists).
  Interventions: Behavioral: ACT in group
- Improved Treatment as usual by General practitioner (Active Comparator): Patients assigned to this arm will receive treatment as usual by their General Practitioner in the Primary Care center. To enhance treatment, investigators participating in the trial will receive the Guidelines for fibromyalgia treatment in Primary Care handed by Health Service in Aragón.
  Interventions: Behavioral: Improved treatment as usual by General Practitioners

INTERVENTIONS:
Behavioral: ACT in group — A protocol based on the main research studies describing the therapy and adapted for fibromyalgia treatment by our research group will be used. This protocol is available for the investigators. There will be 9 group sessions of 90 minutes duration each. Patients assigned to this arm will be allowed to occasionally take minor analgesics.
  Other Names: Acceptation Committment Therapy in group.
  Arms: ACT in group
Behavioral: Improved treatment as usual by General Practitioners — General practitioners (GPs) will administer treatment as usual to the patients with fibromyalgia. To enhance the intervention, the Clinical Guidelines on the Treatment of Fibromyalgia approved by the Health Services of Aragon will be provided to the GPs.
  Other Names: Improved Treatment as Usual
  Arms: Improved Treatment as usual by General practitioner

SUMMARY:
The main objective is to assess the efficacy of Acceptance & Commitment Therapy (ACT) in group for the treatment of fibromyalgia. The secondary aims are: 1.- To assess the cost-effectiveness of ACT and 2.- To assess the efficacy of ACT in other variables such as anxiety, depression, pain or global function. 3.- To evaluate the usefulness or electroencephalographic cordance as a prognostic variable of the treatment.

HYPOTHESIS: ACT in group is effective for improvement of pain acceptance and other outcome variables (pain, anxiety, depression, global function) in fibromyalgia, and it is cost-effective. Cordance is an useful predictor of treatment efficacy in these patients.

DESIGN: Multicentre, randomized, controlled study, with parallel groups, and a 6-month follow-up period. Participants will be randomly allocated to one of two conditions: 1.- Group Acceptation & Commitment Therapy or 2.- Treatment as usual by his general practitioner. Patients diagnosed of fibromyalgia, according to the American College of Rheumatology, will be recruited in primary care. Assuming an alpha=0.05 and p=80%, using two tails, and calculating 5% of refusals, it will be necessary a sample size of 55 patients for each group of patients.

DETAILED DESCRIPTION:
The main outcome will be pain acceptance. Other outcome measures will be global function (assessed with the Fibromyalgia Impact Questionnaire, FIQ), cost-effectiveness (evaluated by the Client Service Receipt Inventory, CSRI) and electroencephalographic cordance. The mediating variables included are anxiety and depression (assessed with the Hospital Anxiety and Depression scale, HADS) and pain (measured with an analog visual scale). A psychiatric interview will be administered to the participants to diagnose Posttraumatic Stress Disorder. Statistical analysis will be carried out for intention to treat, and using the method Last Observation Carried Forward. A Repeated Measures Mixed Model will be used to study the main outcome. All calculations will be made with two tails and a significance of 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-65 year old
2. Discontinuation drug treatment 7 days before the start of the trial
3. Not having received psychological treatment previously or at least in the last 2 years
4. Ability to understand Spanish
5. Given consent to participate in the study

Exclusion Criteria:

1. Age: <18 year old and > 65 year old
2. Clinical or psychological disease that, at investigator's opinion, can interfere the psychological examination or the adherence to psychotherapy (dementia, alcohol or drug abuse, psychosis, severe personality disorder)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-07 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
GLOBAL FUNCTION | At baseline
  GLOBAL FUNCTION is assessed with the Fibromyalgia Impact Questionnaire (FIQ), a 10-item self report questionnaire to evaluate health status of patients with fibromyalgia. The Spanish version will be used.
GLOBAL FUNCTION | At month 3
  GLOBAL FUNCTION is assessed with the Fibromyalgia Impact Questionnaire (FIQ), a 10-item self report questionnaire to evaluate health status of patients with fibromyalgia. The Spanish version will be used.
GLOBAL FUNCTION | At month 6
  GLOBAL FUNCTION is assessed with the Fibromyalgia Impact Questionnaire (FIQ), a 10-item self report questionnaire to evaluate health status of patients with fibromyalgia. The Spanish version will be used.
GLOBAL FUNCTION | At month 9
  GLOBAL FUNCTION is assessed with the Fibromyalgia Impact Questionnaire (FIQ), a 10-item self report questionnaire to evaluate health status of patients with fibromyalgia. The Spanish version will be used.

SECONDARY OUTCOMES:
DEMOGRAPHIC AND CLINICAL DATA | At Baseline
  It has been designed a questionnaire to collect demographic data (sex, age, marital status, education level, job, work disability) and clinical data (psychiatric medical history, disease duration, main symptoms, medical comorbidity etc)
PAIN CATASTROPHIZING | At Baseline
  It is described as a negative and exaggerated reaction towards painful stimulus. It is measured with the Pain Catastrophizing Scale that allows investigators to discriminate 3 sub-scales: rumination, magnification and helplessness. The Spanish validation of this scale will be used.
ANXIETY AND DEPRESSION | At Baseline
  They will be evaluated with the Hospital Anxiety and Depression Scale (HADS), a scale to detect anxiety and depression in people with medical diseases such as fibromyalgia. It is a 14-item self report scale in which items are scored in a Likert scale from 1 to 4. It includes 2 subscales: anxiety and depression, scored independently. The HADS has been validated in Spanish.
PSYCHIATRIC DIAGNOSIS | At baseline
  The Standardized Polyvalent Psychiatric Interview (SPPI) will be used. It is a psychiatric interview developed by our research group to assess psychiatric morbidity in primary care. It allows the use of different diagnosis criteria like DSM-IV and ICD-10. The Posttraumatic stress disorder will be assessed specifically as it has been shown to be related to a worse prognosis in fibromyalgia.
PAIN | At baseline
  It will be assessed with The Analogue Visual Pain Scale. Pain is self-reported by the patient in a visual analogue scale from 0 (pain absence) to 100 (the worst pain anyone can ever imagine)
COST-EFFECTIVENESS ANALYSIS | At Baseline
  COST-EFFECTIVENESS ANALYSIS: Includes a) Drug profile, and b) Services.
PAIN ACCEPTANCE | At Baseline
  Acceptance is related to a better adaptation to pain response, no matter the influence of outcomes such as depression, pain intensity or anxiety. The Chronic Pain Acceptance Questionnaire will be used. This outcome will be measured with the Spanish version validated by our research group.
CORDANCE | At baseline
  CORDANCE: the Fast Fourier Transform (FFT) will be applied to artefact-free electroencephalogram activity segments to calculate absolute and relative powers for each electrode.
PAIN CATASTROPHIZING | At month 3
  It is described as a negative and exaggerated reaction towards painful stimulus. It is measured with the Pain Catastrophizing Scale that allows investigators to discriminate 3 sub-scales: rumination, magnification and helplessness. The Spanish validation of this scale will be used.
PAIN CATASTROPHIZING | At month 6
  It is described as a negative and exaggerated reaction towards painful stimulus. It is measured with the Pain Catastrophizing Scale that allows investigators to discriminate 3 sub-scales: rumination, magnification and helplessness. The Spanish validation of this scale will be used.
ANXIETY AND DEPRESSION | At month 3
  They will be evaluated with the Hospital Anxiety and Depression Scale (HADS), a scale to detect anxiety and depression in people with medical diseases such as fibromyalgia. It is a 14-item self report scale in which items are scored in a Likert scale from 1 to 4. It includes 2 subscales: anxiety and depression, scored independently. The HADS has been validated in Spanish.
ANXIETY AND DEPRESSION | At month 6
  They will be evaluated with the Hospital Anxiety and Depression Scale (HADS), a scale to detect anxiety and depression in people with medical diseases such as fibromyalgia. It is a 14-item self report scale in which items are scored in a Likert scale from 1 to 4. It includes 2 subscales: anxiety and depression, scored independently. The HADS has been validated in Spanish.
PAIN | At month 3
  It will be assessed with The Analogue Visual Pain Scale. Pain is self-reported by the patient in a visual analogue scale from 0 (pain absence) to 100 (the worst pain anyone can ever imagine)
PAIN | At month 6
  It will be assessed with The Analogue Visual Pain Scale. Pain is self-reported by the patient in a visual analogue scale from 0 (pain absence) to 100 (the worst pain anyone can ever imagine)
COST-EFFECTIVENESS ANALYSIS | At month 3
  COST-EFFECTIVENESS ANALYSIS: Includes a) Drug profile, and b) Services.
COST-EFFECTIVENESS ANALYSIS | At month 6
  COST-EFFECTIVENESS ANALYSIS: Includes a) Drug profile, and b) Services.
COST-EFFECTIVENESS ANALYSIS | At month 9
  COST-EFFECTIVENESS ANALYSIS: Includes a) Drug profile, and b) Services.
PAIN ACCEPTANCE | At month 3
  Acceptance is related to a better adaptation to pain response, no matter the influence of outcomes such as depression, pain intensity or anxiety. The Chronic Pain Acceptance Questionnaire will be used. This outcome will be measured with the Spanish version validated by our research group.
PAIN ACCEPTANCE | At month 6
  Acceptance is related to a better adaptation to pain response, no matter the influence of outcomes such as depression, pain intensity or anxiety. The Chronic Pain Acceptance Questionnaire will be used. This outcome will be measured with the Spanish version validated by our research group.
PAIN ACCEPTANCE | At month 9
  Acceptance is related to a better adaptation to pain response, no matter the influence of outcomes such as depression, pain intensity or anxiety. The Chronic Pain Acceptance Questionnaire will be used. This outcome will be measured with the Spanish version validated by our research group.
CORDANCE | At month 3
  CORDANCE: the Fast Fourier Transform (FFT) will be applied to artefact-free electroencephalogram activity segments to calculate absolute and relative powers for each electrode.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Alda, Principal Investigator — Hospital Miguel Servet
Locations (1):
- Mental Health Unit, Primary Care Center "Torrero-La Paz", Zaragoza, Zaragoza, Spain

REFERENCES:
- [Background] Wolfe F, Smythe HA, Yunus MB, Bennett RM, Bombardier C, Goldenberg DL, Tugwell P, Campbell SM, Abeles M, Clark P, et al. The American College of Rheumatology 1990 Criteria for the Classification of Fibromyalgia. Report of the Multicenter Criteria Committee. Arthritis Rheum. 1990 Feb;33(2):160-72. doi: 10.1002/art.1780330203. PMID 2306288
- [Background] Garcia-Campayo J, Sanz-Carrillo C, Baringo T, Ceballos C. SPECT scan in somatization disorder patients: an exploratory study of eleven cases. Aust N Z J Psychiatry. 2001 Jun;35(3):359-63. doi: 10.1046/j.1440-1614.2001.00909.x. PMID 11437810
- [Background] Cook DB, Lange G, Ciccone DS, Liu WC, Steffener J, Natelson BH. Functional imaging of pain in patients with primary fibromyalgia. J Rheumatol. 2004 Feb;31(2):364-78. PMID 14760810
- [Background] McCracken LM. Learning to live with the pain: acceptance of pain predicts adjustment in persons with chronic pain. Pain. 1998 Jan;74(1):21-27. doi: 10.1016/S0304-3959(97)00146-2. PMID 9514556
- [Background] McCracken LM, Vowles KE, Eccleston C. Acceptance of chronic pain: component analysis and a revised assessment method. Pain. 2004 Jan;107(1-2):159-66. doi: 10.1016/j.pain.2003.10.012. PMID 14715402
- [Background] Leuchter AF, Cook IA, Lufkin RB, Dunkin J, Newton TF, Cummings JL, Mackey JK, Walter DO. Cordance: a new method for assessment of cerebral perfusion and metabolism using quantitative electroencephalography. Neuroimage. 1994 Jun;1(3):208-19. doi: 10.1006/nimg.1994.1006. PMID 9343572
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Garcia-Campayo J, Pascual A, Alda M, Marzo J, Magallon R, Fortes S. The Spanish version of the FibroFatigue Scale: validation of a questionnaire for the observer's assessment of fibromyalgia and chronic fatigue syndrome. Gen Hosp Psychiatry. 2006 Mar-Apr;28(2):154-60. doi: 10.1016/j.genhosppsych.2005.12.001. PMID 16516066
- [Background] Garcia-Campayo J, Pascual A, Alda M, Ramirez MTG. Coping with fibromialgia: usefulness of the Chronic Pain Coping Inventory-42. Pain. 2007 Nov;132 Suppl 1:S68-S76. doi: 10.1016/j.pain.2007.02.013. Epub 2007 Apr 2. PMID 17400387
- [Background] Garcia Campayo J, Rodero B, Alda M, Sobradiel N, Montero J, Moreno S. [Validation of the Spanish version of the Pain Catastrophizing Scale in fibromyalgia]. Med Clin (Barc). 2008 Oct 18;131(13):487-92. doi: 10.1157/13127277. Spanish. PMID 19007576
- [Background] Garcia-Campayo J, Serrano-Blanco A, Rodero B, Magallon R, Alda M, Andres E, Luciano JV, del Hoyo YL. Effectiveness of the psychological and pharmacological treatment of catastrophization in patients with fibromyalgia: a randomized controlled trial. Trials. 2009 Apr 23;10:24. doi: 10.1186/1745-6215-10-24. PMID 19389246
- [Background] Garcia-Campayo J, Magdalena J, Magallon R, Fernandez-Garcia E, Salas M, Andres E. A meta-analysis of the efficacy of fibromyalgia treatment according to level of care. Arthritis Res Ther. 2008;10(4):R81. doi: 10.1186/ar2455. Epub 2008 Jul 15. PMID 18627602